CLINICAL TRIAL: NCT05997056
Title: A Phase 2 Multi-center, Open-label, Single Arm Study of Nab-sirolimus in Patients With Well-differentiated Neuroendocrine Tumors (NETs) of the Gastrointestinal Tract, Lung, or Pancreas Who Have Not Received Prior Treatment With mTOR Inhibitors
Brief Title: Trial of Nab-sirolimus in Patients With Well-differentiated Neuroendocrine Tumors (NETs) of the Gastrointestinal Tract, Lung, or Pancreas Who Have Not Received Prior Treatment With mTOR Inhibitors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NET-202
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Neuroendocrine Tumors; NET; Pancreatic Neuroendocrine Tumor; Gastrointestinal Neuroendocrine Tumor; Pulmonary Neuroendocrine Tumor
Keywords: FYARRO; nab-sirolimus; ABI-009; Neuroendocrine Tumors; NET; Pancreatic Neuroendocrine Tumor; Gastrointestinal Neuroendocrine Tumor; Pulmonary Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors; Adenoma, Islet Cell; Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- neuroendocrine tumors (Experimental): Patients with well-differentiated neuroendocrine tumors of the gastrointestinal tract, lung, or pancreas.
  Interventions: Drug: nab-sirolimus

INTERVENTIONS:
Drug: nab-sirolimus — Prospective phase 2 single arm, open-label, multi-institutional study to determine the efficacy and safety prospective of nab-sirolimus administered by IV infusion
  Other Names: ABI-009

SUMMARY:
A Phase 2 multi-center, open-label, single arm study of nab-sirolimus in patients with well-differentiated neuroendocrine tumors (NETs) of the gastrointestinal tract, lung, or pancreas who have not received prior treatment with mTOR inhibitors

DETAILED DESCRIPTION:
This is a prospective phase 2 single arm, open-label, multi-institutional study to determine the efficacy and safety prospective of nab-sirolimus and patients with functional or non-functional, well-differentiated, locally advanced unresectable in metastatic NETs of the GI tract, lung, or pancreas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with functional or non-functional, well-differentiated, locally advanced unresectable or metastatic NETs of the GI tract, lung, or pancreas who have received 2 or less prior lines of therapy excluding somatostatin analogs
2. Patients with functional NETs may enroll if:

   1. the patient has been on a stable dose of an somatostatin analogs for ≥12 weeks and
   2. the patient has experienced disease progression while on stable somatostatin analogs dose
3. Patients must have 1 or more measurable target lesions by RECIST v1.1
4. Age: 18 years or older
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 or Karnofsky Performance Status (KPS) ≥80
6. Adequate liver function:

   1. Total bilirubin ≤1.5 × upper limit of normal (ULN) (unless due to Gilbert's syndrome or attributable to liver metastases, then ≤3 × ULN)
   2. Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤2.5 × ULN (≤5 × ULN if attributable to liver metastases)
7. Adequate renal function: creatinine clearance ≥30 mL/min, Cockcroft-Gault creatinine clearance = ((140-age) × weight[kg]) / (72 × serum creatinine [mL/min]) × 0.85, if female.
8. Adequate hematologic parameters:

   1. Absolute neutrophil count (ANC) ≥1.0 × 10^9/L (growth factor support allowed)
   2. Platelet count ≥100,000/mm^3 (100 × 10^9/L) (transfusion and/or growth factor support allowed)
   3. Hemoglobin ≥8.0 g/dL (transfusion and/or growth factor support allowed)
9. Fasting serum triglyceride must be ≤300 mg/dL; fasting serum cholesterol must be less than or equal to 350 mg/dL
10. Minimum of 4 weeks since any major surgery, completion of radiation, and adequately recovered from the acute toxicities of any prior therapy, including neuropathy, to Grade ≤1
11. Male or non-pregnant and non-breastfeeding female:

    1. Females of childbearing potential must agree to use effective contraception or abstinence without interruption from 28 days prior to starting study medication throughout 3 months after last dose of study medication and have a negative serum pregnancy test (beta human chorionic gonadotropin [β-hCG]) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the EOS treatment. A second form of birth control is required even if she has had a tubal ligation.
    2. Male patients must agree not to donate sperm and must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study and throughout 3 months after last dose of study medication. A second form of birth control is required even if he has undergone a successful vasectomy.
    3. Sexual abstinence is considered a highly effective contraceptive method only if defined as refraining from heterosexual intercourse from 28 days prior to starting study medication throughout 3 months after last dose of study medication. The reliability of sexual abstinence should be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the patient.
12. The patient or the patient's legal guardian(s) understand(s) and sign(s) the informed consent
13. Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures
14. Patients with a known history of human immunodeficiency virus (HIV) infection are eligible if:

    1. There has been no acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection in 12 months prior to enrollment.
    2. The patient has been receiving an antiretroviral therapy regimen for ≥4 weeks and the HIV viral load is <400 copies/mL prior to enrollment.
    3. Antiretroviral therapy regimen does not include strong cytochrome (CYP)3A4 inhibitors or inducers

Exclusion Criteria:

1. Prior treatment with mTOR inhibitors including nab-sirolimus

   Note: Patients who have previously received locoregional or liver-directed therapies (radiofrequency or microwave ablation, transarterial chemoembolization, etc.) are eligible to enroll in the study.
2. Patients with functional NETs who are experiencing uncontrolled symptoms attributed to hormones and other vasoactive substances secreted by the tumor
3. Patients with inactivating TSC1 or TSC2 alterations (based on tissue or liquid NGS)
4. Severe (Grade ≥3) ongoing infection requiring parenteral or oral anti-infective treatment, either ongoing or completed ≤7 days prior to enrollment
5. Patients who have any severe and/or uncontrolled medical or psychiatric conditions or other conditions that could affect their participation including:

   1. Known or suspected brain metastases
   2. Severe heart disease defined as unstable angina pectoris, NYHA Class III or IV congestive heart failure, myocardial infarction ≤6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
   3. Severe lung disease defined as a diffusing capacity for carbon monoxide that is ≤50% of normal predicted value and/or an O2 saturation ≤88% at rest on room air

      (Note: Spirometry and pulmonary function tests are not required to be performed unless clinically indicated.)
   4. Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
   5. A history of malignancies other than the one under treatment unless the patient is disease-free for more than 5 years from diagnosis. Controlled non-melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer, certain low-grade hematologic malignancies (eg, chronic lymphocytic leukemia, follicular lymphoma, etc), or other adequately treated carcinoma in situ may be eligible, after discussion with the medical monitor.
   6. Uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg)
   7. Patients with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension
   8. Active Hepatitis B and/or Hepatitis C infection and detectable viral load despite antiviral therapy.
6. Required use of concomitant medications with strong CYP3A4 interactions (induction or inhibition) should be discontinued (strong inhibitors include ketoconazole, itraconazole, voriconazole, erythromycin, clarithromycin, telithromycin; strong inducers include rifampin and rifabutin). These agents must be discontinued prior to first dose of nab-sirolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-05-09 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of nab-sirolimus | 12 Months
  Objective Response Rate (ORR), defined as the proportion of patients with best overall response (BOR) of confirmed partial response (PR) or complete response (CR) from the time of study treatment initiation until progression of disease (PD) as determined by the Investigator using RECIST v1.1

SECONDARY OUTCOMES:
Incidence and severity of treatment | 12 Months
  Incidence and severity of treatment-emergent and treatment-related adverse events (AEs) as assessed by NCI CTCAE v5.0
Duration of response | 12 Months
  Determined for patients with BOR of confirmed CR or PR defined as time from scan first showing response by RECIST v1.1 to PD or death
Disease control rate | 12 Months
  BOR of confirmed CR or PR (either of any duration) or stable disease (SD) ≥12 weeks by RECISTv1.1 following study treatment initiation
Time to response | 12 Months
  Time from first dose of study medication to initial measurement of CR or PR, where CR or PR is subsequently confirmed by RECIST v1.1
Progression-free survival | 12 Months
  Number of months from study treatment initiation to the date of disease progression or death due to any cause
Overall survival | 24 Months
  Number of months from study treatment initiation to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Willis Navarro, MD, Study Director — Aadi Bioscience
Locations (4):
- United States (4):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Texas Oncology, Dallas, Texas
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No